CLINICAL TRIAL: NCT05287776
Title: The Effect of Narrow Band UVB on E-cadherin and Integrin Alpha v Beta 1 in Non-segmental Vitiligo: A Novel Proposed Mechanism
Brief Title: E-cadherin and Integrin Alpha v Beta 1 in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer of dermatology, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EcadVitiligo
Record Dates: First submitted 2021-09-22; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15 patients with vitiligo subjected to NB-UVB (Experimental): Patients will be subjected to NB-UVB sessions 3 times weekly. The UVB dosing scheme in the patients receiving only NB-UVB treatment entailed initial dosing at 0.5 J/cm2 with increasing increments by 0.3 J/cm 2 every other session until faint erythema occurs.
  Interventions: Device: Narrow band UVB

INTERVENTIONS:
Device: Narrow band UVB — Narrow band UVB emitting UVB at wavelength 311nm

SUMMARY:
The purpose of this clinical trial is to study the effect of Narrow Band UVB on E-cadherin and integrin alpha v beta 1 as representatives of adhesion molecules in non-segmental vitiligo in a trial to verify a novel proposed mechanism of Narrow Band UVB. Additionally, specific melanocyte marker (Melan A) will be done to settle the localization of adhesion molecules in relation to melanocytes.

ELIGIBILITY:
Inclusion Criteria:

* All clinically diagnosed cases of non-segmental vitiligo .
* Patients with VIDA +1 or more (new/expanding lesions active in time period of 6-12 months ago) will be included in the trial. Activity of vitiligo will be evaluated through Vitiligo Disease Activity (VIDA) Score.

Exclusion Criteria:

* Patients who have stable disease at the time of study i.e. no progression of existing disease or appearance of new lesions in the last six months.
* Patients receiving treatment for vitiligo 3 months prior to the study.
* Patients with contraindications for phototherapy.
* Patients with current/history of any systemic and/or dermatological diseases affecting the immune system as autoimmune diseases and malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Melanocyte marker (Melan A) for staining of melanocytes | 4 months
  Immunohistochemistry and image analysis Data were obtained using Leica Quinn software with Olympus BX40 microscope and Panasonic camera Measurements were taken in 5 non-overlapping high power fields.
E-cadherin expression as a cell adhesion molecule between melanocytes and keratinocytes | 4 months
  Immunohistochemistry and image analysis Data were obtained using Leica Quinn software with Olympus BX40 microscope and Panasonic camera Measurements were taken in 5 non-overlapping high power fields.
Integrin alpha v beta 1 expression as a cell adhesion molecule between melanocytes and keratinocytes | 4 months
  Immunohistochemistry and image analysis Data were obtained using Leica Quinn software with Olympus BX40 microscope and Panasonic camera Measurements were taken in 5 non-overlapping high power fields.

SECONDARY OUTCOMES:
Vitiligo Area and severity index (VASI) | 4 months
  Minimum value is 0, maximum value is 100 Higher scores mean worse outcome

OTHER OUTCOMES:
Vitiligo Disease Activity score (VIDA) | 4 months
  Minimum value -1, maximum value 4 Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy university hospital, Faulty of medicine,Cairo university, Cairo, El Manial, Egypt